CLINICAL TRIAL: NCT06566469
Title: Effect of Dexmedetomidine-esketamine Combined Nasal Administration on Emergence Delirium in Elderly Patients After Surgery: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Dexmedetomidine-esketamine Combined Nasal Administration and Emergence Delirium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-405
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Older Patients; Nasal Administration; Dexmedetomidine; Esketamine; General Anesthesia; Emergence Delirium
Keywords: Older patients; Nasal administration; Dexmedetomidine; Esketamine; General anesthesia; Emergence delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined dexmedetomidine-esketamine (Experimental): A mixture of dexmedetomidine 0.5 µg/kg and esketamine 0.2 mg/kg is administered via nasal spray at 20:30 pm the day before surgery and at 07:30 am and 20:30 pm the day of surgery.
  Interventions: Drug: Dexmedetomidine; Drug: Esketamine
- Normal saline (Placebo Comparator): Placebo (normal saline) at the same volume is administered via nasal spray at 20:30 pm the day before surgery and at 07:30 am and 20:30 pm the day of surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.5 µg/kg is administered via nasal spray at 20:30 pm the day before surgery and at 07:30 am and 20:30 pm the day of surgery.
  Arms: Combined dexmedetomidine-esketamine
Drug: Esketamine — Esketamine 0.2 mg/kg is administered via nasal spray at 20:30 pm the day before surgery and at 07:30 am and 20:30 pm the day of surgery.
  Arms: Combined dexmedetomidine-esketamine
Drug: Normal saline — Normal saline at the same volume is administered via nasal spray at 20:30 pm the day before surgery and at 07:30 am and 20:30 pm the day of surgery.
  Arms: Normal saline

SUMMARY:
Emergence delirium is common in older patients after surgery and associated with worse perioperative outcomes, including increased postoperative delirium. Nasal administrations of both dexmedetomidine and esketamine are approved for medical purposes. Combination of low-dose dexmedetomidine and esketamine has shown some synergic effects in analgesia and anxiolysis. In a recent randomized trial, combined nasal administration of dexmedetomidine and esketamine was more effective in reducing pre-dental anxiety in pediatric patients. The investigators hypothesize that perioperative nasal administration of dexmedetomidine-esketamine combination can reduce the incidence of emergence delirium in older patients after surgery.

DETAILED DESCRIPTION:
Delirium is a common brain dysfunction syndrome in older patients after major surgery. Delirium that occurs after surgery includes emergence delirium and postoperative delirium. Emergence delirium occurred in 17.5% to 37.0% of patients following general anesthesia. The reported incidence of postoperative delirium ranged from 12.0% to 32.9% in older patients after noncardiac surgery. It is well known that the occurrence of postoperative delirium is associated with adverse outcomes. Recent studies found that emergence delirium is also associated with adverse perioperative outcomes, including increased postoperative delirium, more non-delirium complications, longer hospital stay, and higher healthcare costs.

Dexmedetomidine is a highly selective alpha 2-adrenoceptor agonist with sedative, anxiolytic, and analgesic effects. Prophylactic administration of dexmedetomidine preoperatively or intraoperatively has also been shown to reduce the incidence of postoperative delirium. Dexmedetomidine via nasal administration is now widely used for pediatric preoperative sedation. Nasal administration of dexmedetomidine is also used in adults. In a retrospective study, postoperative nasal administration of dexmedetomidine (100 μg) to elderly orthopedic surgical patients improved analgesia and reduced symptoms of agitation. A recent study of patients undergoing gynecologic laparoscopic surgery, night-time dexmedetomidine (1.5 µg/kg) administration by nasal drops from preoperative day 1 to postoperative day 5 improved sleep quality and reduced the incidence of postoperative delirium.

Esketamine is a N-methyl-D-aspartic acid receptor antagonist and has been used as an anesthetic and analgesic. Low-dose intravenous infusion of ketamine is recommended for postoperative analgesia. Esketamine is s-enantiomer of ketamine and twice as potent as ketamine in analgesic potency. Nasal administration of esketamine is approved by FDA for intractable depression in adults. A randomized trial showed that nasal application of esketamine was effective in relieving post-thoracic puncture pain in adult patients without significant adverse effects. And postoperative pain is a common risk factor of emergence delirium and postoperative delirium.

This randomized trial is designed to test the hypothesis that combined nasal administration of dexmedetomidine-esketamine combination may reduce the incidence of emergence delirium in older patients after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 65 years;
2. Scheduled for inpatient elective or semi-elective surgery under general anesthesia, with an expected surgical duration of ≤2 hours;
3. Planned to stay in hospital for at least 1 day after surgery.

Exclusion Criteria:

1. Not suitable for intranasal drug administration due to nasal disease (e.g., rhinitis, nasal polyps, or nasal congestion due to any cause);
2. Preoperative schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, or delirium;
3. Inability to communicate due to coma, severe dementia, or language barrier before surgery;
4. Brain trauma or neurosurgery;
5. Use of sedatives or hypnotics at bedtime during the last month;
6. History of hyperthyroidism or pheochromocytoma;
7. Preoperative left ventricular ejection fraction <30%, or sick sinus node syndrome, severe sinus bradycardia (heart rate <50 beats per minute), or atrioventricular block of degree II or higher without pacemaker, or systolic blood pressure <90 mmHg before enrollment;
8. Severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (receiving dialysis before surgery), or American Society of Anesthesiologists classification ≥ IV;
9. Planned admission to the intensive care unit after surgery;
10. Allergic to dexmedetomidine and/or esketamine, or any other conditions that are considered unsuitable for study participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 340 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Incidence of emergence delirium after surgery | During stay in the post-anesthesia care unit
  Emergence delirium is assessed with the Richmond Agitation Sedation Scale (RASS; scores range from -5 [unarousable] to +4 [combative] and 0 indicates alert and calm) and the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) at 5 and 30 minutes after admission to the post-anesthesia care unit.

SECONDARY OUTCOMES:
Incidence of emergence agitation | During anesthesia emergence in the operating room
  Emergence agitation is assessed with the RASS after surgery from cessation of general anesthesia to leaving operating room. A RASS score ≥+2 at any time is defined as having emergence agitation.
Subjective sleep quality score | The night before surgery and the night of surgery
  Subjective sleep quality is assessed with the Richards-Campbell Sleep Questionnaire (RCSQ). The RCSQ is a self-reported measure that evaluates perception of nighttime sleep in five items, including sleep depth, sleep latency, number of awakenings, returning to sleep, and overall sleep quality. Each item is assessed with a 100 millimeter visual analog scale (score ranges from 0 to 100, with higher scores indicating better sleep quality). The mean score of the five items represents the overall sleep quality.
Incidence of delayed neurocognitive recovery | At 5 days after surgery
  Cognition is assessed with the telephone-Montreal Cognitive Assessment (T-MoCA; score ranges from 0 to 22, with higher score indicating better function). A reducation of T-MoCA score of ≥1 standard deviation (SD) from baseline is defined as having delayed neurocognitive recovery.

OTHER OUTCOMES:
Pain intensity within 24 hours after surgery | Up to 24 hours after surgery
  Pain intensity is assessed with the numeric rating scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) at 5 and 30 minutes on the day of surgery and between 8 and 10 am and 18 and 20 pm on the first day after surgery.
Analgesic use within 24 hours after surgery | Up to 24 hours after surgery
  Includes opioids and non-opioid analgesics.
Incidence of postoperative delirium within 3 days after surgery | Up to 3 days after surgery
  Postoperative delirium is assessed twice daily (8-10 am and 18-20 pm) with the 3-minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) for non-intubated patients or the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) for intubated patients.
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery.
Subjective sleep quality at 30 day after surgery | At 30 days after surgery
  Subjective sleep quality at 30 days is assessed with the Pittsburgh Sleep Quality Index (PSQI). PSQI is a 7-item questionnaire consisting 19 self-rated questions that assesses sleep quality over the last month, each weighted equally on a 0-3 scale; higher scores indicate worse sleep quality
Incidence of postoperative complications within 30 days after surgery | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical events that are deemed harmful and required therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcantonio ER. Postoperative delirium: a 76-year-old woman with delirium following surgery. JAMA. 2012 Jul 4;308(1):73-81. doi: 10.1001/jama.2012.6857. PMID 22669559
- [Background] Silverstein JH, Timberger M, Reich DL, Uysal S. Central nervous system dysfunction after noncardiac surgery and anesthesia in the elderly. Anesthesiology. 2007 Mar;106(3):622-8. doi: 10.1097/00000542-200703000-00026. No abstract available. PMID 17325520
- [Background] Aldecoa C, Bettelli G, Bilotta F, Sanders RD, Audisio R, Borozdina A, Cherubini A, Jones C, Kehlet H, MacLullich A, Radtke F, Riese F, Slooter AJ, Veyckemans F, Kramer S, Neuner B, Weiss B, Spies CD. European Society of Anaesthesiology evidence-based and consensus-based guideline on postoperative delirium. Eur J Anaesthesiol. 2017 Apr;34(4):192-214. doi: 10.1097/EJA.0000000000000594. PMID 28187050
- [Background] Card E, Pandharipande P, Tomes C, Lee C, Wood J, Nelson D, Graves A, Shintani A, Ely EW, Hughes C. Emergence from general anaesthesia and evolution of delirium signs in the post-anaesthesia care unit. Br J Anaesth. 2015 Sep;115(3):411-7. doi: 10.1093/bja/aeu442. Epub 2014 Dec 23. PMID 25540068
- [Background] Hesse S, Kreuzer M, Hight D, Gaskell A, Devari P, Singh D, Taylor NB, Whalin MK, Lee S, Sleigh JW, Garcia PS. Association of electroencephalogram trajectories during emergence from anaesthesia with delirium in the postanaesthesia care unit: an early sign of postoperative complications. Br J Anaesth. 2019 May;122(5):622-634. doi: 10.1016/j.bja.2018.09.016. Epub 2018 Oct 25. PMID 30915984
- [Background] Zhang Y, He ST, Nie B, Li XY, Wang DX. Emergence delirium is associated with increased postoperative delirium in elderly: a prospective observational study. J Anesth. 2020 Oct;34(5):675-687. doi: 10.1007/s00540-020-02805-8. Epub 2020 Jun 7. PMID 32507939
- [Background] Wu J, Gao S, Zhang S, Yu Y, Liu S, Zhang Z, Mei W. Perioperative risk factors for recovery room delirium after elective non-cardiovascular surgery under general anaesthesia. Perioper Med (Lond). 2021 Feb 3;10(1):3. doi: 10.1186/s13741-020-00174-0. PMID 33531068
- [Background] Gu WJ, Zhou JX, Ji RQ, Zhou LY, Wang CM. Incidence, risk factors, and consequences of emergence delirium after elective brain tumor resection. Surgeon. 2022 Oct;20(5):e214-e220. doi: 10.1016/j.surge.2021.09.005. Epub 2021 Nov 12. PMID 34782237
- [Background] Tesfaye Mekonin G, Kelbesa Olika M, Birhanu Wedajo M, Tolasa Badada A, Dukessa Dubiwak A, Tageza Ilala T, Gebre MN. Prevalence of Emergence Delirium and Associated Factors among Older Patients Who Underwent Elective Surgery: A Multicenter Observational Study. Anesthesiol Res Pract. 2022 Sep 9;2022:2711310. doi: 10.1155/2022/2711310. eCollection 2022. PMID 36119120
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844
- [Background] Berian JR, Zhou L, Russell MM, Hornor MA, Cohen ME, Finlayson E, Ko CY, Rosenthal RA, Robinson TN. Postoperative Delirium as a Target for Surgical Quality Improvement. Ann Surg. 2018 Jul;268(1):93-99. doi: 10.1097/SLA.0000000000002436. PMID 28742701
- [Background] Saravana-Bawan B, Warkentin LM, Rucker D, Carr F, Churchill TA, Khadaroo RG. Incidence and predictors of postoperative delirium in the older acute care surgery population: a prospective study. Can J Surg. 2019 Feb 1;62(1):33-38. doi: 10.1503/cjs.016817. PMID 30693744
- [Background] Tawab Saljuqi A, Hanna K, Asmar S, Tang A, Zeeshan M, Gries L, Ditillo M, Kulvatunyou N, Castanon L, Joseph B. Prospective Evaluation of Delirium in Geriatric Patients Undergoing Emergency General Surgery. J Am Coll Surg. 2020 May;230(5):758-765. doi: 10.1016/j.jamcollsurg.2020.01.029. Epub 2020 Feb 21. PMID 32088308
- [Background] Silva AR, Regueira P, Albuquerque E, Baldeiras I, Cardoso AL, Santana I, Cerejeira J. Estimates of Geriatric Delirium Frequency in Noncardiac Surgeries and Its Evaluation Across the Years: A Systematic Review and Meta-analysis. J Am Med Dir Assoc. 2021 Mar;22(3):613-620.e9. doi: 10.1016/j.jamda.2020.08.017. Epub 2020 Oct 1. PMID 33011097
- [Background] Igwe EO, Nealon J, O'Shaughnessy P, Bowden A, Chang HR, Ho MH, Montayre J, Montgomery A, Rolls K, Chou KR, Chen KH, Traynor V, Smerdely P. Incidence of postoperative delirium in older adults undergoing surgical procedures: A systematic literature review and meta-analysis. Worldviews Evid Based Nurs. 2023 Jun;20(3):220-237. doi: 10.1111/wvn.12649. Epub 2023 May 2. PMID 37128953
- [Background] Bao L, Liu T, Zhang Z, Pan Q, Wang L, Fan G, Li Z, Yin Y. The prediction of postoperative delirium with the preoperative bispectral index in older aged patients: a cohort study. Aging Clin Exp Res. 2023 Jul;35(7):1531-1539. doi: 10.1007/s40520-023-02408-9. Epub 2023 May 19. PMID 37204755
- [Background] Liu XH, Zhang QF, Liu Y, Lu QW, Wu JH, Gao XH, Chen ZY. Risk factors associated with postoperative delirium in elderly patients undergoing hip surgery. Front Psychiatry. 2023 Oct 19;14:1288117. doi: 10.3389/fpsyt.2023.1288117. eCollection 2023. PMID 37928911
- [Background] Gleason LJ, Schmitt EM, Kosar CM, Tabloski P, Saczynski JS, Robinson T, Cooper Z, Rogers SO Jr, Jones RN, Marcantonio ER, Inouye SK. Effect of Delirium and Other Major Complications on Outcomes After Elective Surgery in Older Adults. JAMA Surg. 2015 Dec;150(12):1134-40. doi: 10.1001/jamasurg.2015.2606. PMID 26352694
- [Background] Ha A, Krasnow RE, Mossanen M, Nagle R, Hshieh TT, Rudolph JL, Chang SL. A contemporary population-based analysis of the incidence, cost, and outcomes of postoperative delirium following major urologic cancer surgeries. Urol Oncol. 2018 Jul;36(7):341.e15-341.e22. doi: 10.1016/j.urolonc.2018.04.012. Epub 2018 May 24. PMID 29801992
- [Background] Park EA, Kim MY. Postoperative Delirium is Associated with Negative Outcomes and Long-Term Mortality in Elderly Koreans: A Retrospective Observational Study. Medicina (Kaunas). 2019 Sep 20;55(10):618. doi: 10.3390/medicina55100618. PMID 31547219
- [Background] Oberai T, Woodman R, Laver K, Crotty M, Kerkhoffs G, Jaarsma R. Is delirium associated with negative outcomes in older patients with hip fracture: analysis of the 4904 patients 2017-2018 from the Australian and New Zealand hip fracture registry. ANZ J Surg. 2022 Jan;92(1-2):200-205. doi: 10.1111/ans.17421. Epub 2021 Dec 13. PMID 34904334
- [Background] Ma X, Chu H, Han K, Shao Q, Yu Y, Jia S, Wang D, Wang Z, Zhou Y. Postoperative delirium after transcatheter aortic valve replacement: An updated systematic review and meta-analysis. J Am Geriatr Soc. 2023 Feb;71(2):646-660. doi: 10.1111/jgs.18104. Epub 2022 Nov 23. PMID 36419366
- [Background] Crocker E, Beggs T, Hassan A, Denault A, Lamarche Y, Bagshaw S, Elmi-Sarabi M, Hiebert B, Macdonald K, Giles-Smith L, Tangri N, Arora RC. Long-Term Effects of Postoperative Delirium in Patients Undergoing Cardiac Operation: A Systematic Review. Ann Thorac Surg. 2016 Oct;102(4):1391-9. doi: 10.1016/j.athoracsur.2016.04.071. Epub 2016 Jun 22. PMID 27344279
- [Background] Shi Z, Mei X, Li C, Chen Y, Zheng H, Wu Y, Zheng H, Liu L, Marcantonio ER, Xie Z, Shen Y. Postoperative Delirium Is Associated with Long-term Decline in Activities of Daily Living. Anesthesiology. 2019 Sep;131(3):492-500. doi: 10.1097/ALN.0000000000002849. PMID 31335550
- [Background] Goldberg TE, Chen C, Wang Y, Jung E, Swanson A, Ing C, Garcia PS, Whittington RA, Moitra V. Association of Delirium With Long-term Cognitive Decline: A Meta-analysis. JAMA Neurol. 2020 Nov 1;77(11):1373-1381. doi: 10.1001/jamaneurol.2020.2273. PMID 32658246
- [Background] Huang H, Li H, Zhang X, Shi G, Xu M, Ru X, Chen Y, Patel MB, Ely EW, Lin S, Zhang G, Zhou J. Association of postoperative delirium with cognitive outcomes: A meta-analysis. J Clin Anesth. 2021 Dec;75:110496. doi: 10.1016/j.jclinane.2021.110496. Epub 2021 Sep 2. PMID 34482263
- [Background] Pereira JV, Aung Thein MZ, Nitchingham A, Caplan GA. Delirium in older adults is associated with development of new dementia: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2021 Jul;36(7):993-1003. doi: 10.1002/gps.5508. Epub 2021 Feb 27. PMID 33638566
- [Background] Mohanty S, Gillio A, Lindroth H, Ortiz D, Holler E, Azar J, Boustani M, Zarzaur B. Major Surgery and Long Term Cognitive Outcomes: The Effect of Postoperative Delirium on Dementia in the Year Following Discharge. J Surg Res. 2022 Feb;270:327-334. doi: 10.1016/j.jss.2021.08.043. Epub 2021 Oct 29. PMID 34731730
- [Background] Moskowitz EE, Overbey DM, Jones TS, Jones EL, Arcomano TR, Moore JT, Robinson TN. Post-operative delirium is associated with increased 5-year mortality. Am J Surg. 2017 Dec;214(6):1036-1038. doi: 10.1016/j.amjsurg.2017.08.034. Epub 2017 Sep 20. PMID 28947274
- [Background] Yokoyama C, Yoshitnai K, Ogata S, Fukushima S, Matsuda H. Effect of postoperative delirium after cardiovascular surgery on 5-year mortality. JA Clin Rep. 2023 Oct 13;9(1):66. doi: 10.1186/s40981-023-00658-0. PMID 37831211
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Niu JY, Yang N, Tao QY, He Y, Hou YB, Ning RD, Yu JM. Effect of Different Administration Routes of Dexmedetomidine on Postoperative Delirium in Elderly Patients Undergoing Elective Spinal Surgery: A Prospective Randomized Double-Blinded Controlled Trial. Anesth Analg. 2023 Jun 1;136(6):1075-1083. doi: 10.1213/ANE.0000000000006464. Epub 2023 Apr 14. PMID 37058430
- [Background] Ghazaly HF, Hemaida TS, Zaher ZZ, Elkhodary OM, Hammad SS. A pre-anesthetic bolus of ketamine versus dexmedetomidine for prevention of postoperative delirium in elderly patients undergoing emergency surgery: a randomized, double-blinded, placebo-controlled study. BMC Anesthesiol. 2023 Dec 11;23(1):407. doi: 10.1186/s12871-023-02367-8. PMID 38082227
- [Background] Li S, Li R, Li M, Cui Q, Zhang X, Ma T, Wang D, Zeng M, Li H, Bao Z, Peng Y, Sessler DI. Dexmedetomidine administration during brain tumour resection for prevention of postoperative delirium: a randomised trial. Br J Anaesth. 2023 Feb;130(2):e307-e316. doi: 10.1016/j.bja.2022.10.041. Epub 2022 Dec 13. PMID 36517290
- [Background] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Background] Li A, Yuen VM, Goulay-Dufay S, Sheng Y, Standing JF, Kwok PCL, Leung MKM, Leung AS, Wong ICK, Irwin MG. Pharmacokinetic and pharmacodynamic study of intranasal and intravenous dexmedetomidine. Br J Anaesth. 2018 May;120(5):960-968. doi: 10.1016/j.bja.2017.11.100. Epub 2018 Feb 2. PMID 29661413
- [Background] Uusalo P, Seppanen SM, Jarvisalo MJ. Feasibility of Intranasal Dexmedetomidine in Treatment of Postoperative Restlessness, Agitation, and Pain in Geriatric Orthopedic Patients. Drugs Aging. 2021 May;38(5):441-450. doi: 10.1007/s40266-021-00846-6. Epub 2021 Mar 16. PMID 33728561
- [Background] He J, Zhang X, Li C, Fu B, Huang Y, Li H. Dexmedetomidine nasal administration improves perioperative sleep quality and neurocognitive deficits in elderly patients undergoing general anesthesia. BMC Anesthesiol. 2024 Jan 30;24(1):42. doi: 10.1186/s12871-024-02417-9. PMID 38291398
- [Background] Barrett W, Buxhoeveden M, Dhillon S. Ketamine: a versatile tool for anesthesia and analgesia. Curr Opin Anaesthesiol. 2020 Oct;33(5):633-638. doi: 10.1097/ACO.0000000000000916. PMID 32826629
- [Background] Wolff K, Winstock AR. Ketamine : from medicine to misuse. CNS Drugs. 2006;20(3):199-218. doi: 10.2165/00023210-200620030-00003. PMID 16529526
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Pfenninger EG, Durieux ME, Himmelseher S. Cognitive impairment after small-dose ketamine isomers in comparison to equianalgesic racemic ketamine in human volunteers. Anesthesiology. 2002 Feb;96(2):357-66. doi: 10.1097/00000542-200202000-00022. PMID 11818769
- [Background] Sapkota A, Khurshid H, Qureshi IA, Jahan N, Went TR, Sultan W, Alfonso M. Efficacy and Safety of Intranasal Esketamine in Treatment-Resistant Depression in Adults: A Systematic Review. Cureus. 2021 Aug 21;13(8):e17352. doi: 10.7759/cureus.17352. eCollection 2021 Aug. PMID 34447651
- [Background] Xu J, Jian J, Zhang Y, Wu J, Qiu Y. The efficacy of nasal administration of esketamine in patients having moderate-to-severe pain after preoperative CT-guided needle localization: a randomized, double-blind, placebo-controlled trial. Front Med (Lausanne). 2024 Apr 9;11:1344160. doi: 10.3389/fmed.2024.1344160. eCollection 2024. PMID 38654836
- [Background] He M, Zhu Z, Jiang M, Liu X, Wu R, Zhou J, Chen X, Liu C. Risk Factors for Postanesthetic Emergence Delirium in Adults: A Systematic Review and Meta-analysis. J Neurosurg Anesthesiol. 2024 Jul 1;36(3):190-200. doi: 10.1097/ANA.0000000000000942. Epub 2023 Nov 2. PMID 37916963
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Sica R, Wilson JM, Kim EJ, Culley DJ, Meints SM, Schreiber KL. The Relationship of Postoperative Pain and Opioid Consumption to Postoperative Delirium After Spine Surgery. J Pain Res. 2023 Jan 28;16:287-294. doi: 10.2147/JPR.S380616. eCollection 2023. PMID 36744116
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Background] Xing F, Zhang TT, Yang Z, Qu M, Shi X, Li Y, Li Y, Zhang W, Wang Z, Xing N. Comparison of dexmedetomidine and a dexmedetomidine-esketamine combination for reducing dental anxiety in preschool children undergoing dental treatment under general anesthesia: A randomized controlled trial. J Affect Disord. 2024 Feb 15;347:569-575. doi: 10.1016/j.jad.2023.12.011. Epub 2023 Dec 6. PMID 38065480
- [Background] Huge V, Lauchart M, Magerl W, Schelling G, Beyer A, Thieme D, Azad SC. Effects of low-dose intranasal (S)-ketamine in patients with neuropathic pain. Eur J Pain. 2010 Apr;14(4):387-94. doi: 10.1016/j.ejpain.2009.08.002. Epub 2009 Sep 3. PMID 19733106
- [Background] Chen LX, Ji DH, Zhang F, Li JH, Cui L, Bai CJ, Liu H, Liang Y. Richards-Campbell sleep questionnaire: psychometric properties of Chinese critically ill patients. Nurs Crit Care. 2019 Nov;24(6):362-368. doi: 10.1111/nicc.12357. Epub 2018 Jul 30. PMID 30062842
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162